CLINICAL TRIAL: NCT03108495
Title: A Phase 2, Multicenter Study to Evaluate the Efficacy and Safety Using Autologous Tumor Infiltrating Lymphocytes (LN-145) in Patients With Recurrent, Metastatic or Persistent Cervical Carcinoma
Brief Title: Study of LN-145, Autologous Tumor Infiltrating Lymphocytes in the Treatment of Patients With Cervical Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After reviewing available safety and efficacy data to date, Iovance concluded the study reached the required number of events for evaluation of study endpoints.
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-145-04; 2024-510634-41-00 (EU CTIS Number)
Record Dates: First submitted 2017-03-27; First posted 2017-04-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Carcinoma
Keywords: LN-145; Cell Therapy; Autologous Adoptive Cell Transfer; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; Tumor Infiltrating Lymphocytes; TIL; IL-2; Pembrolizumab
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Toll-Like Receptor 1; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 LN-145 monotherapy (Experimental): Post-NMA lymphodepletion, patients are infused with their autologous TIL (LN-145) followed by IL-2 administration.
  Interventions: Biological: LN-145
- Cohort 2 LN-145 monotherapy (Experimental): Patients previously treated with an antiprogrammed cell death protein-1 (PD-1) or anti-programmed death-ligand 1 (PD-L1) checkpoint inhibitor: Post-NMA lymphodepletion, patients are infused with their autologous TIL (LN-145) followed by IL-2 administration.
  Interventions: Biological: LN-145
- Cohort 3 - Combination Arm (TIL + Pembrolizumab) - US Only (Experimental): Patients will be administered with pembrolizumab, followed by NMA lymphodepletion, then infused with their autologous TIL (LN-145) followed by pembrolizumab every 3 or 6 weeks post IL-2 administration up to 24 months.
  Interventions: Biological: LN-145 + pembrolizumab
- Cohort 4 - Non-enrolling Cohort (Experimental): Cohort includes patient population not meeting inclusion criteria in cohort 1 and 2. Post-NMA lymphodepletion, patients are infused with their autologous TIL (LN-145) followed by IL-2 administration.
  Interventions: Biological: LN-145
- Cohort 5 Retreatment Cohort (Experimental): Patients who have been previously treated with LN-145 may be given a second treatment with TIL.
  Interventions: Biological: LN-145

INTERVENTIONS:
Biological: LN-145 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes.
  Other Names: TIL, autologous tumor infiltrating lymphocytes
  Arms: Cohort 1 LN-145 monotherapy; Cohort 2 LN-145 monotherapy; Cohort 4 - Non-enrolling Cohort; Cohort 5 Retreatment Cohort
Biological: LN-145 + pembrolizumab — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. The first dose of anti-PD-1 immunotherapy will be administered following tumor resection.
  Other Names: TIL, autologous tumor infiltrating lymphocytes; pembrolizumab (anti-PD-1 immunotherapy)
  Arms: Cohort 3 - Combination Arm (TIL + Pembrolizumab) - US Only

SUMMARY:
Prospective, multicenter, single-arm, open label, interventional study evaluating adoptive cell therapy (ACT) with autologous tumor infiltrating lymphocytes (TIL) infusion (LN-145) followed by IL-2 after a non-myeloablative (NMA) lymphodepletion preparative regimen for the treatment of patients with recurrent, metastatic, or persistent cervical carcinoma

DETAILED DESCRIPTION:
LN-145 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, as originally developed by the NCI, for the treatment of patients with recurrent, metastatic, or persistent cervical carcinoma. The cell transfer therapy used in this study involves patients receiving a NMA lymphocyte depleting preparative regimen, followed by infusion of autologous TIL followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, patients must meet ALL of the following criteria prior to participation:

1. Must be ≥ 18 years of age at the time of consent. Enrollment of patients > 70 years of age may be allowed after consultation with the Medical Monitor.
2. Must have recurrent, metastatic, or persistent squamous cell carcinoma (SCC), adenosquamous carcinoma (ASC), or adenocarcinoma (AC) of the cervix that is not amenable to curative treatment with surgery and/or radiation therapy.
3. At least one resectable lesion (or aggregate of lesions resected) of a minimum 1.5 cm in diameter post-resection to generate TIL; surgical removal with minimal morbidity (defined as any procedure for which expected hospitalization is ≤ 3 days)
4. At least one measurable target lesion, as defined by RECIST v1.1.
5. Cohort 1 and Cohort 2: Progression during or following at least one, but no more than three, prior systemic chemotherapeutic treatments for recurrent, metastatic, or persistent cervical carcinoma

   * A line of systemic therapy is defined as any chemotherapy or multiple-agent chemotherapy regimen that was administered for recurrent, metastatic, or persistent SCC, ASC, or AC of the cervix.
   * A bevacizumab and chemotherapy combination is encouraged as a prior line of treatment.
   * Neither chemoradiation, nor chemotherapy in the neoadjuvant or adjuvant settings are considered as a prior line of systemic therapy.

   Cohort 2: Must also have previously received treatment with a checkpoint inhibitor (ie, PD-1, PD-L1]) in the setting of recurrent, metastatic, or persistent disease either as monotherapy or in combination (eg, in combination with chemotherapy or another immune agent)

   Cohort 3 (United States only): Must have not received any therapies other than prior chemoradiation or surgery for loco-regional disease
6. Any prior therapy directed at the malignant tumor, including chemotherapy, biologic/targeted agents, and immunologic agents must be discontinued at least 28 days prior to tumor resection.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Must have adequate organ function.
9. Patient has no evidence of any active viral, bacterial, or fungal infection requiring ongoing systemic treatment. Patients must be seronegative for the human immunodeficiency virus (HIV). Patients with acute or chronic hepatitis infections may be enrolled if the viral load by nucleic acid amplification test (NAAT) is undetectable with/without active treatment
10. Patients of childbearing potential must be willing to take the appropriate precaution to avoid pregnancy for the duration of the study and practice an approved, highly effective method of birth control during treatment and for 12 months after receiving the last protocol-related therapy.
11. Prior to study Enrollment (tumor resection), patient must have documentation of radiological disease progression after the most recent therapy

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for participation in this study:

1. Patients who have received an organ allograft or prior cell transfer therapy except for prior LN-145 therapy in the setting of re-treatment only.
2. Patients who require ongoing systemic steroid therapy (> 10 mg/day of prednisone or other steroid equivalent dose).
3. Patients who currently have prior therapy-related toxicities Grade > 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0; except for peripheral neuropathy, alopecia, or vitiligo prior to Enrollment (tumor resection).
4. . Patients who have a history of hypersensitivity to any component or excipient of LN-145 or other study drugs:

   • NMA-LD preparative regimen (cyclophosphamide, mesna, and fludarabine)
5. Patients who have active systemic infections, coagulation disorders, or other active major medical illness(es) of the cardiovascular, respiratory, or immune system, including evidence in the medical history of urinary tract obstruction, a positive cardiac stress test, myocardial infarction, cardiac arrhythmia, obstructive or restrictive pulmonary disease, or other conditions that in the opinion of the Investigator would increase the risk of participation.
6. Patients with symptomatic and/or untreated brain metastases (of any size and any number)

   • Patients with definitively treated brain metastases may be considered for Enrollment, and must be stable for ≥ 14 days prior to beginning the NMA-LD preparative regimen
7. Patients who have any form of primary immunodeficiency (such as severe combined immunodeficiency [SCID] or acquired immunodeficiency syndrome [AIDS])
8. Patients who have a diagnosis of end-stage renal disorder requiring hemodialysis
9. Patients who have a left ventricular ejection fraction (LVEF) < 45% or who are New York Heart Association (NYHA) Class 2 or higher.
10. Patients who have a documented forced expiratory volume in 1 second (FEV1) of ≤ 60%
11. Patients who have had another primary malignancy within the previous 3 years (except for curatively treated localized malignancy that has not required treatment for > 1 year, and in the judgement of the Investigator, does not pose a significant risk of recurrence including, but not limited to, non-melanoma skin cancer or bladder cancer)
12. Patients who are of the following protected classes will be excluded, including:

    * Pregnant, parturient, or breastfeeding women
    * Persons who are hospitalized without consent or those deprived of liberty because of a judiciary or administrative decision
    * Patients with a legal protection measure or a person who cannot express his/her consent
    * Patients in emergency situations who cannot consent to the study
13. Patients who have received a live or attenuated vaccine within 28 days prior to beginning the NMA-LD preparative regimen
14. Patients whose cancer requires immediate attention or who would otherwise suffer a disadvantage by participating in this study
15. Cohort 1 and Cohort 3: Patients who have received prior treatment with immunotherapy (eg, PD-1, PD-L1, or anti-cytotoxic T lymphocyte-associated antigen-4 [CTLA-4] antibodies)
16. Patients who have Grade ≥ 2 hemorrhage within 14 days prior to Enrollment (tumor resection)
17. Cohort 3: Patients may not have active or prior documented autoimmune or inflammatory disorders (including pneumonitis, inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 210 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Cohort 1 and 2: Objective Response Rate | Up to 60 months
  To evaluate the efficacy of LN-145 in patients with recurrent, metastatic, or persistent cervical carcinoma based on the objective response rate (ORR) as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Cohort 3: Adverse Events | Up to 60 months
  To characterize the safety profile of LN-145 in combination with pembrolizumab in patients with recurrent, metastatic, or persistent cervical carcinoma as assessed by incidence of adverse events.
Cohort 4: Efficacy and Adverse Events | Up to 60 months
  To explore the efficacy and safety profile of LN-145 in previously enrolled patients with recurrent, metastatic, or persistent cervical carcinoma
Cohort 5: Efficacy and Adverse Events | Up to 60 months
  To explore the efficacy and safety profile of LN-145 in re-treated patients with recurrent, metastatic, or persistent cervical carcinoma

SECONDARY OUTCOMES:
Cohort 1 and 2: Duration of Response | Up to 60 months
  To evaluate the efficacy parameters of LN-145 in patients with recurrent, metastatic, or persistent cervical carcinoma by assessing duration of response (DOR) as assessed by the Investigator per RECIST v1.1
Cohort 1 and 2: Disease Control Rate | Up to 60 months
  To evaluate the efficacy parameters of LN-145 in patients with recurrent, metastatic, or persistent cervical carcinoma by assessing disease control rate (DCR) as assessed by the Investigator per RECIST v1.1
Cohort 1 and 2: Progression-Free Survival | Up to 60 months
  To evaluate the efficacy parameters of LN-145 in patients with recurrent, metastatic, or persistent cervical carcinoma by assessing progression-free survival (PFS) as assessed by the Investigator per RECIST v1.1
Cohort 1 and 2: Overall Survival | Up to 60 months
  To evaluate overall survival (OS) in patients with recurrent, metastatic, or persistent cervical carcinoma
Cohort 1 and 2: Adverse Events | Up to 60 months
  To characterize the safety profile of LN-145 in patients with recurrent, metastatic, or persistent cervical carcinoma as assessed by incidence of adverse events
Cohort 3: Objective Response Rate | Up to 60 months
  To evaluate the efficacy of LN-145 in combination with pembrolizumab in patients with recurrent, metastatic, or persistent cervical carcinoma based on the objective response rate (ORR) as assessed by the Investigator per RECIST v1.1
Cohort 3: Duration of Response | Up to 60 months
  To evaluate the efficacy of LN-145 in combination with pembrolizumab in patients with recurrent, metastatic, or persistent cervical carcinoma by assessing duration of response (DOR) as assessed by the Investigator per RECIST v1.1.
Cohort 3: Disease Control Rate | Up to 60 months
  To evaluate the efficacy of LN-145 in combination with pembrolizumab in patients with recurrent, metastatic, or persistent cervical carcinoma by assessing disease control rate (DCR) as assessed by the Investigator per RECIST v1.1.
Cohort 3: Progression-Free Survival | Up to 60 months
  To evaluate the efficacy of LN-145 in combination with pembrolizumab in patients with recurrent, metastatic, or persistent cervical carcinoma by assessing progression-free survival (PFS) as assessed by the Investigator per RECIST v1.1.
Cohort 3: Overall Survival | Up to 60 months
  To evaluate overall survival (OS) in patients with recurrent, metastatic, or persistent cervical carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Medical Monitor, Study Director — Iovance Biotherapeutics, Inc.
Locations (43):
- United States (24):
  - St. Joseph's Hospital and Medical Center Center For Women's Health, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - University of Florida Health Cancer Center, Orlando, Florida
  - University of South Florida H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers University, Newark, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Allegheny Health, Pittsburgh, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Avera Medical Group Oncology, Sioux Falls, South Dakota
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- France (3):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Léon Bérard, Lyon
  - Gustave Roussy Cancer Campus, Villejuif
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
- Istituto Europeo di Oncologia, Miano, Milano, Italy
- Academisch Medisch Centrum, Amsterdam, AZ, Netherlands
- Spain (5):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Institut Català d'Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
- Switzerland (2):
  - Inselspital, Bern
  - Centre Hospitalier Universitaire Vaudois Lausanne - Centre Pluridisciplinaire d'Oncologie, Lausanne
- United Kingdom (5):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Sarah Cannon Research Institute London, London, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - NHS Greater Glasgow and Clyde, Glasgow, Scotland
  - Guy's & St.Thomas NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No